CLINICAL TRIAL: NCT04579302
Title: Evaluation of the Effect of Serratus Anterior Block and Erector Spinae Block on Postoperative Analgesia in Thoracic Surgeries
Brief Title: Serratus Anterior Block and Erector Spinae Block in Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AP2007-50105
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Analgesia
Keywords: Serratus anterior block; Erector spinae block; Postoperative analgesia
MeSH Terms: interventions — Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- serratus anterior block (Experimental): serratus anterior block with 20 ml bupivacaine
  Interventions: Procedure: Serratus anterior block (SAB); Drug: Bupivacaine
- erector spinae block (Experimental): erector spinae block with 20 ml bupivacaine
  Interventions: Procedure: Erector spinae block; Drug: Bupivacaine
- control group (Sham Comparator): sham block with 20 ml saline
  Interventions: Drug: Saline (as a placebo)

INTERVENTIONS:
Procedure: Serratus anterior block (SAB) — Patients will receive a sonar guided serratus anterior plane block with 20 ml of bupivacaine 0.5%
  Other Names: SAB group
  Arms: serratus anterior block
Procedure: Erector spinae block — Patients will receive a sonar-guided erector spinae plane block with 20 ml of bupivacaine 0.5%
  Other Names: ESB group
  Arms: erector spinae block
Drug: Saline (as a placebo) — Patients will receive a sham block with 20 ml saline (as a placebo)
  Arms: control group
Drug: Bupivacaine — bupivacaine
  Arms: erector spinae block; serratus anterior block

SUMMARY:
90 patients scheduled for thoracic cancer surgeries, allocated in 3 groups for serratus anterior block and erector spinae block and control group. during anaesthesia:total intraoperative fentanyl required will be recorded. After surgery, all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded.

DETAILED DESCRIPTION:
90 patients scheduled for thoracic cancer surgeries, allocated in 3 groups for serratus anterior block (SAB) and erector spinae block (ESB) and control group. During anaesthesia: total intraoperative fentanyl required will be recorded. After surgery, all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded. Other secondary outcomes are: numerical rating scales and postoperative pulmonary functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class II physical status (American Society of Anaesthesiologists) ,
* Age between 18-70 years,
* Scheduled for thoracic cancer surgery

Exclusion Criteria:

* Patient refusal.
* Local infection at the site of the block.
* Cardiac dysfunction (ejection fraction <45%).
* Significant respiratory disorders.
* Preexisting neurological or psychiatric disease.
* Allergy to one of the study drugs.
* Pregnancy.
* Coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
total morphine consumption in first postoperative 24 hours | first 24 postoperative hours
  the amount of morphine required to relieve pain will be recorded

SECONDARY OUTCOMES:
intraoperative fentanyl requirement | during anaesthesia
  the amount of fentanyl required during anaesthesia will be recorded
numerical rating scale | the first 24 postoperative hours
  numerical rating scale (from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain) will be recorded in different time intervals during the first 24 hours after surgery
pulmonary functions | 24 hours after surgery
  FVC and FEV1 will be recorded at 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Hassan, MS, Principal Investigator — National Cancer Institute - Vairo University - Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No